CLINICAL TRIAL: NCT00264758
Title: Frequent Hemodialysis Network: Daily Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: beck-daily; 5U01DK066597 (NIH)
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: End Stage Renal Disease
Keywords: randomized controlled clinical trial; hemodialysis; end stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional hemodialysis (Active Comparator): Three times per week in-center hemodialysis
  Interventions: Device: Conventional hemodialysis
- Frequent hemodialysis (Experimental): Six times per week in-center hemodialysis
  Interventions: Device: Frequent hemodialysis

INTERVENTIONS:
Device: Conventional hemodialysis — Three times per week in-center hemodialysis
  Arms: Conventional hemodialysis
Device: Frequent hemodialysis — Six times per week in-center hemodialysis
  Arms: Frequent hemodialysis

SUMMARY:
The Frequent Hemodialysis Network (FHN) Daily Trial is a randomized controlled trial recruiting subjects from dialysis units associated with designated Clinical Centers in the U.S. and Canada and followed for 1 year. Subjects will be randomized to either conventional hemodialysis Daily HD delivered for at least 2.5 hours (typically 3 to 4 hours), 3 days per week, or to more frequent hemodialysis delivered for 1.5 - 2.75 hours, 6 days per week. The study has two co-primary outcomes: 1) a composite of mortality with the change over 12 months in left ventricular mass by magnetic resonance imaging, and 2) a composite of mortality with the change over 12 months in the SF-36 RAND physical health composite (PHC) quality of life scale.

DETAILED DESCRIPTION:
This trial is a randomized controlled trial recruiting subjects from dialysis units associated with designated Clinical Centers in the U.S. and Canada. A total of 250 ESRD patients receiving in-center HD will be randomized to continue with conventional HD, 3 days per week (control group), or switch to daily HD, 6 days per week (intervention group). Subjects will be treated and followed for 12 months. Two co-primary outcomes are designated: 1) a composite of mortality with the change over 12 months in left ventricular mass, and 2) a composite of mortality with the change over 12 months in the SF-36 RAND physical health composite. In addition, main secondary outcomes have been designated for each of seven outcome domains: 1) cardiovascular structure and function (change in LV mass), 2) health-related quality of life/physical function (change in the PHC), 3) depression/burden of illness (change in Beck Depression Inventory), 4) nutrition (change in serum albumin), 5) cognitive function (change in the Trail Making Test B), 6) mineral metabolism (change in average predialysis serum phosphorus), and 7) clinical events (rate of non-access hospitalization or death). Hypertension and anemia are also main outcome domains, but without designation of single first priority outcomes.

The objectives of this study are the following:

Feasibility:

1. To determine the feasibility of recruiting and retaining patients in a randomized trial of six times per week in-center daily HD versus conventional three times per week in-center HD.
2. To determine patient adherence with and acceptance of in-center daily HD, and to identify reasons for discontinuation from or nonadherence with the therapy.

   Safety:
3. To determine the safety of in-center daily HD with a particular focus on vascular access events and participant burden.

   Efficacy:
4. To evaluate the efficacy of in-center daily HD compared to conventional three times per week HD on two co-primary outcomes: i) a composite of mortality with the change over 12 months in left ventricular mass by magnetic resonance imaging (MRI), and ii) a composite of mortality with the change over 12 months in the SF-36 RAND physical health composite score (PHC).
5. To determine the effect of in-center daily HD on nine secondary outcome domains: i) cardiovascular structure and function, ii) health-related quality of life and physical function, iii) depression/burden of illness, iv) nutrition and inflammation, v) cognitive function, vi) mineral metabolism, vii) clinical events, viii) hypertension, and ix) anemia.

   Characterization of the Intervention
6. To better understand the complex therapy of in-center daily HD, by evaluating solute clearance, treatment times, volume removal, and non-dialytic factors such as differences in the frequency of medical surveillance and treatment.

   Implementation:
7. To determine the feasibility of implementing in-center daily HD in practice, by evaluating barriers to implementation such as the incremental cost of daily HD compared to 3 times per week conventional HD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with end stage renal disease requiring chronic renal replacement therapy
2. Age 13 years or greater
3. Achieved mean eKt/V of > 1.0 on at least two baseline sessions
4. Weight 30 kg or greater

Exclusion Criteria:

1. Residual renal urea clearance > 3 mL/min per 35 L.
2. Expectation that native kidneys will recover
3. Vascular access being used for HD is a non-tunneled catheter
4. Inability to come for in-center 6 days a week, including inability to arrange adequate transportation
5. History of poor adherence to thrice weekly HD
6. Medical conditions that would prevent the subject from performing the cardiac MRI procedure (e.g., inability to remain still for the procedure, a metallic object in the body, including cardiac pacemaker, inner ear (cochlear) implant, brain aneurysm clips, mechanical heart valves, recently placed artificial joints, and older vascular stents)
7. Unable to verbally communicate in English or Spanish
8. Requires HD > 3 times per week due to medical co-morbidity (such as, but not limited to: systemic oxalosis, or requiring total parenteral nutrition). Occasional ultrafiltration on a fourth day per week is not an exclusion criterion.
9. Currently on daily or nocturnal HD, or less than 3 months since the subject discontinued daily or nocturnal HD
10. Scheduled for living donor kidney transplant, change to peritoneal dialysis, home HD, or plans to relocate to another center within the next 14 months
11. Expected geographic unavailability at a participating HD unit for > 2 consecutive weeks or > 4 weeks total during the next 14 months (excluding unavailability due to hospitalizations) (frequent HD subjects who leave for vacation may resort back to conventional HD during these time periods)
12. Less than 3 months since the patient returned to HD after acute rejection resulting in allograft failure
13. Currently in acute or chronic care hospital
14. Life expectancy < 6 months
15. A medical history that might limit the subject's ability to take trial treatments for the 12 month duration of the study, including: currently receiving chemo or radiotherapy for a malignant neoplastic disease other than localized non-melanoma skin cancer, active systemic infection (including tuberculosis, disseminated fungal infection, active AIDS but not HIV, and cirrhosis with encephalopathy)
16. Current pregnancy, or actively planning to become pregnant in the next 12 months
17. Contraindication to heparin, including allergy or heparin induced thrombocytopenia
18. Current use of investigational drugs or participation in another clinical trial that contradicts or interferes with the therapies or measured outcomes in this trial
19. Unable or unwilling to follow the study protocol for any reason (including mental incompetence)
20. Unable or unwilling to provide informed consent or sign IRB-approved consent form

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2006-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
a composite of mortality with the change over 12 months in left ventricular mass | 12 months
a composite of mortality with the change over 12 months in the SF-36 RAND physical health composite. | 12 months

SECONDARY OUTCOMES:
cardiovascular structure and function (change in LV mass) | 12 months
health-related quality of life/physical function (change in the PHC) | 12 months
depression/burden of illness (change in Beck Depression Inventory) | 12 months
nutrition (change in serum albumin) | 12 months
cognitive function (change in the Trail Making Test B) | 12 months
mineral metabolism (change in average predialysis serum phosphorus) | 12 months
clinical events (rate of non-access hospitalization or death) | 12 months
hypertension | 12 months
anemia | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul W. Eggers, Ph.D., Study Director — NIDDK, NIH; Glenn Chertow, M.D., Principal Investigator — University of California, San Francisco; Nathan W. Levin, M.D., Principal Investigator — Renal Research Institute; Gerald J. Beck, Ph.D., Principal Investigator — The Cleveland Clinic; Alan S. Kliger, M.D., Study Chair — Yale New Haven Health System
Locations (2):
- United States (2):
  - University of California at San Francisco - Core center plus other centers in California and Texas, San Francisco, California
  - Renal Research Institute - Core center plus other centers in U.S. and Canada, New York, New York

REFERENCES:
- [Background] Suri RS, Garg AX, Chertow GM, Levin NW, Rocco MV, Greene T, Beck GJ, Gassman JJ, Eggers PW, Star RA, Ornt DB, Kliger AS; Frequent Hemodialysis Network Trial Group. Frequent Hemodialysis Network (FHN) randomized trials: study design. Kidney Int. 2007 Feb;71(4):349-59. doi: 10.1038/sj.ki.5002032. Epub 2006 Dec 13. PMID 17164834
- [Background] Kliger AS; Frequent Hemodialysis Network Study Group. High-frequency hemodialysis: rationale for randomized clinical trials. Clin J Am Soc Nephrol. 2007 Mar;2(2):390-2. doi: 10.2215/CJN.03110906. Epub 2006 Dec 20. No abstract available. PMID 17699439
- [Result] Rocco MV, Larive B, Eggers PW, Beck GJ, Chertow GM, Levin NW, Kliger AS; FHN Trial Group. Baseline characteristics of participants in the Frequent Hemodialysis Network (FHN) daily and nocturnal trials. Am J Kidney Dis. 2011 Jan;57(1):90-100. doi: 10.1053/j.ajkd.2010.08.024. Epub 2010 Nov 30. PMID 21122961
- [Result] FHN Trial Group; Chertow GM, Levin NW, Beck GJ, Depner TA, Eggers PW, Gassman JJ, Gorodetskaya I, Greene T, James S, Larive B, Lindsay RM, Mehta RL, Miller B, Ornt DB, Rajagopalan S, Rastogi A, Rocco MV, Schiller B, Sergeyeva O, Schulman G, Ting GO, Unruh ML, Star RA, Kliger AS. In-center hemodialysis six times per week versus three times per week. N Engl J Med. 2010 Dec 9;363(24):2287-300. doi: 10.1056/NEJMoa1001593. Epub 2010 Nov 20. PMID 21091062
- [Result] Daugirdas JT, Greene T, Rocco MV, Kaysen GA, Depner TA, Levin NW, Chertow GM, Ornt DB, Raimann JG, Larive B, Kliger AS; FHN Trial Group. Effect of frequent hemodialysis on residual kidney function. Kidney Int. 2013 May;83(5):949-58. doi: 10.1038/ki.2012.457. Epub 2013 Jan 23. PMID 23344474
- [Result] Chan CT, Chertow GM, Daugirdas JT, Greene TH, Kotanko P, Larive B, Pierratos A, Stokes JB; Frequent Hemodialysis Network Daily Trial Group. Effects of daily hemodialysis on heart rate variability: results from the Frequent Hemodialysis Network (FHN) Daily Trial. Nephrol Dial Transplant. 2014 Jan;29(1):168-78. doi: 10.1093/ndt/gft212. Epub 2013 Sep 26. PMID 24078335
- [Derived] Moloney BM, Chertow GM, Mc Causland FR. Association of Diabetes with Heart Rate Variability during Hemodialysis: Insights from the Frequent Hemodialysis Network Daily Trial. Kidney360. 2025 Mar 13;6(7):1127-1134. doi: 10.34067/KID.0000000765. PMID 40080097
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553
- [Derived] Chan CT, Kaysen GA, Beck GJ, Li M, Lo JC, Rocco MV, Kliger AS; FHN Trials. The effect of frequent hemodialysis on matrix metalloproteinases, their tissue inhibitors, and FGF23: Implications for blood pressure and left ventricular mass modification in the Frequent Hemodialysis Network trials. Hemodial Int. 2020 Apr;24(2):162-174. doi: 10.1111/hdi.12807. Epub 2019 Dec 11. PMID 31826326
- [Derived] Chan CT, Kaysen GA, Beck GJ, Li M, Lo J, Rocco MV, Kliger AS; FHN Trials. Changes in Biomarker Profile and Left Ventricular Hypertrophy Regression: Results from the Frequent Hemodialysis Network Trials. Am J Nephrol. 2018;47(3):208-217. doi: 10.1159/000488003. Epub 2018 Apr 5. PMID 29621747
- [Derived] Lo JC, Beck GJ, Kaysen GA, Chan CT, Kliger AS, Rocco MV, Li M, Chertow GM; FHN Study. Thyroid function in end stage renal disease and effects of frequent hemodialysis. Hemodial Int. 2017 Oct;21(4):534-541. doi: 10.1111/hdi.12527. Epub 2017 Mar 16. PMID 28301073
- [Derived] Garg AX, Suri RS, Eggers P, Finkelstein FO, Greene T, Kimmel PL, Kliger AS, Larive B, Lindsay RM, Pierratos A, Unruh M, Chertow GM; Frequent Hemodialysis Network Trial Investigators. Patients receiving frequent hemodialysis have better health-related quality of life compared to patients receiving conventional hemodialysis. Kidney Int. 2017 Mar;91(3):746-754. doi: 10.1016/j.kint.2016.10.033. Epub 2017 Jan 13. PMID 28094031
- [Derived] Raimann JG, Abbas SR, Liu L, Zhu F, Larive B, Kotanko P, Levin NW, Kaysen GA; FHN Trial. Agreement of single- and multi-frequency bioimpedance measurements in hemodialysis patients: an ancillary study of the Frequent Hemodialysis Network Daily Trial. Nephron Clin Pract. 2014;128(1-2):115-26. doi: 10.1159/000366447. Epub 2014 Nov 7. PMID 25402657
- [Derived] Chan CT, Greene T, Chertow GM, Kliger AS, Stokes JB, Beck GJ, Daugirdas JT, Kotanko P, Larive B, Levin NW, Mehta RL, Rocco M, Sanz J, Yang PC, Rajagopalan S; Frequent Hemodialysis Network Trial Group. Effects of frequent hemodialysis on ventricular volumes and left ventricular remodeling. Clin J Am Soc Nephrol. 2013 Dec;8(12):2106-16. doi: 10.2215/CJN.03280313. Epub 2013 Aug 22. PMID 23970131
- [Derived] Unruh ML, Larive B, Chertow GM, Eggers PW, Garg AX, Gassman J, Tarallo M, Finkelstein FO, Kimmel PL; FHN Trials Group. Effects of 6-times-weekly versus 3-times-weekly hemodialysis on depressive symptoms and self-reported mental health: Frequent Hemodialysis Network (FHN) Trials. Am J Kidney Dis. 2013 May;61(5):748-58. doi: 10.1053/j.ajkd.2012.11.047. Epub 2013 Jan 15. PMID 23332990
- [Derived] Kurella Tamura M, Unruh ML, Nissenson AR, Larive B, Eggers PW, Gassman J, Mehta RL, Kliger AS, Stokes JB; Frequent Hemodialysis Network (FHN) Trial Group. Effect of more frequent hemodialysis on cognitive function in the frequent hemodialysis network trials. Am J Kidney Dis. 2013 Feb;61(2):228-37. doi: 10.1053/j.ajkd.2012.09.009. Epub 2012 Nov 11. PMID 23149295
- [Derived] Hall YN, Larive B, Painter P, Kaysen GA, Lindsay RM, Nissenson AR, Unruh ML, Rocco MV, Chertow GM; Frequent Hemodialysis Network Trial Group. Effects of six versus three times per week hemodialysis on physical performance, health, and functioning: Frequent Hemodialysis Network (FHN) randomized trials. Clin J Am Soc Nephrol. 2012 May;7(5):782-94. doi: 10.2215/CJN.10601011. Epub 2012 Mar 15. PMID 22422538
- [Derived] Chan CT, Greene T, Chertow GM, Kliger AS, Stokes JB, Beck GJ, Daugirdas JT, Kotanko P, Larive B, Levin NW, Mehta RL, Rocco M, Sanz J, Schiller BM, Yang PC, Rajagopalan S; Frequent Hemodialysis Network (FHN) Trial Group. Determinants of left ventricular mass in patients on hemodialysis: Frequent Hemodialysis Network (FHN) Trials. Circ Cardiovasc Imaging. 2012 Mar;5(2):251-61. doi: 10.1161/CIRCIMAGING.111.969923. Epub 2012 Feb 23. PMID 22360996
- [Derived] Chan CT, Levin NW, Chertow GM, Larive B, Schulman G, Kotanko P; Frequent Hemodialysis Network Daily Trial Group. Determinants of cardiac autonomic dysfunction in ESRD. Clin J Am Soc Nephrol. 2010 Oct;5(10):1821-7. doi: 10.2215/CJN.03080410. Epub 2010 Jul 8. PMID 20616163
- [Derived] Greene T, Daugirdas JT, Depner TA, Gotch F, Kuhlman M; Frequent Hemodialysis Network Study Group; National Institute of Diabetes and Digestive and Kidney Diseases; National Institutes of Health. Solute clearances and fluid removal in the frequent hemodialysis network trials. Am J Kidney Dis. 2009 May;53(5):835-44. doi: 10.1053/j.ajkd.2008.12.039. Epub 2009 Apr 1. PMID 19339093